CLINICAL TRIAL: NCT05196412
Title: Screening of Cardiac Arrhythmias With Wrist-worn Aino ECG Cardiac Monitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseOn Oy (Industry)
Collaborators: TAYS Sydänkeskus Oy (Unknown); Atostek Oy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AinoScreening
Record Dates: First submitted 2021-11-18; First posted 2022-01-19 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Arrhythmias, Cardiac; Atrial Fibrillation
Keywords: Wearable; Wrist-worn
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main study group (Experimental): Normal subjects of at least 65 years of age
  Interventions: Device: PulseOn Arrhythmia Monitor device
- Endurance athlete group (Experimental): Group consists of active endurance athletes of at least 50 years of age
  Interventions: Device: PulseOn Arrhythmia Monitor device

INTERVENTIONS:
Device: PulseOn Arrhythmia Monitor device — Wearing of the wrist device for a period of two weeks

SUMMARY:
The study investigates the performance pf PulseOn Arrhythmia Monitor System that includes a wrist-worn device, which combines continuous optical heartbeat interval monitoring and intermittent ECG measurement, and a data management system used by healthcare professionals for data observation, in the detection of previously undiagnosed cardiac arrhythmias, especially atrial fibrillation.

DETAILED DESCRIPTION:
The study consists of monitoring voluntary subjects with PulseOn Arrhythmia Monitoring System for the period of two weeks. The subjects are recruited mainly through newspaper advertisements. The study is executed in Tampere and Helsinki areas, Finland.

During the two week monitoring time, the subjects are instructed to wear the wrist device continuously, except when taking the device off e.g. for going to sauna or swimming, and for charging. The subjects are instructed to perform a 35-second ECG measurement (recording) in three cases:

1. Scheduled recording four times a day
2. In case of suspecting arrhythmic event, i.e. feeling symptoms
3. In case the wrist device instructs to perform a recording by vibrating and showing an LED light

The data collected in the study is analysed post-hoc. In the post-hoc analysis, the cardiac rhythm assessed automatically from the ECG measurements is visually confirmed by a cardiologist.

ELIGIBILITY:
Inclusion Criteria for the main study group:

* At least 65 years of age
* Self-assessed ability to use the study devices
* Ability to give informed consent
* Volunteering for the study

Inclusion criteria for the active endurance athlete group:

* Minimum of 10 years of active training of endurance sport (e.g. long distance running, skiing, cycling, triathlon…) and currently an average amount of training of at least 10 hours a week.
* Age: ≥ 50 years
* Self-assessed ability to use the study devices
* Ability to give informed consent
* Volunteering for the study

Exclusion Criteria for both groups:

* Cardiac pacemaker
* Earlier diagnosis of atrial fibrillation
* Inability to give informed consent
* Denial

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-05-22 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance improvement with continuous optical measurement | Duration of patient measurement, i.e. two weeks
  Percentual improvement in the performance of detecting previously undiagnosed atrial fibrillation in the study population by the continuous PPG-based heartbeat interval monitoring when compared with relying only on scheduled and symptom -based ECG measurements. Cardiac rhythm assessed by a cardiologist from the ECG measurements that are made as a result of PPG-based arrhythmia notifications is compared with rhythm assessments made only from the scheduled and symptom-based ECG measurements. It is evaluated whether more subjects can be diagnosed having atrial fibrillation with the help of continuous PPG-based rhythm monitoring.
Validation of the clinical performance of PulseOn Arrhythmia Monitor System in general population by showing the adequacy of the obtained ECG data for clinical decision making. | Duration of patient measurement, i.e. two weeks
  Data recorded by the study subjects during the two-week study time is assessed by a cardiologist and subjects are classified as having: "no observed arrhythmias", "atrial fibrillation episode(s)", "other potential arrhythmia", or "unconfident assessment" (due to the quality or lack of data). The percentage of "unconfident assessment" shall be less than 20% of the subjects.
Validation of the clinical performance of PulseOn Arrhythmia Monitor System in general population by showing sufficient patient convenience for using the device for the intended duration of two weeks | Duration of patient measurement, i.e. two weeks
  The feedback from the subjects should show at least grade 3 in a scale of 1-5 for the "comfortability of using the wrist device".

SECONDARY OUTCOMES:
Showing the benefit of the combined wrist-worn PPG and ECG solution in detecting other cardiac arrhythmias than atrial fibrillation. | Duration of patient measurement, i.e. two weeks
  The visual ECG-based rhythm annotation made by a cardiologist is compared with simultaneous PPG-algorithm alarm state. The incidence of notifications for other arrhythmias than atrial fibrilation is reported.
Evaluation of the necessity of performing scheduled ECG measurements in addition to ECG measurements triggered by PPG-based arrhythmia notifications for detecting atrial fibrillation. | Duration of patient measurement, i.e. two weeks
  Evaluation is done by comparing the atrial fibrillation detection outcome when considering only the PPG-triggered and symptom-based ECG measurements or when considering also the scheduled ECG measurements. The outcome parameter is the number of subjects that would have been left undetected if the scheduled ECG measurements were not taken.
Feedback about the usability of the evaluated solution from study subjects. | At the end of the 2-week measurement period
  Feedback questions in scale of 1-5 and open-ended feedback. Easiness of use of the wrist device, understandability of the user interface, suitability of the user materials, and unobtrusiveness.
Feedback about the usability of the evaluated solution from study personnel. | At the end of the study i.e. the end of 2022.
  Feedback questions in scale of 1-5 and open-ended feedback. Easiness of use of the data management service, suitability of the user materials.
Quality of the measured ECG signals | Duration of patient measurement, i.e. two weeks
  Percentage of the ECG measurements classified as inadequate quality for rhythm assessment either an ECG analysis algorithm or by a doctor.
Assessment of the subjects' adherence in using the solution. | Duration of patient measurement, i.e. two weeks
  Analysis of how well the participants will follow the study protocol and do the participants register their ECG in correlation with the wrist device notification. The outcome parameter is the percentage of scheduled and PPG-based notifications to take an ECG measurement and the variation of the percentage between the subjects.
Benefit of optical measurement for the speed of detecting atrial fibrillation | Duration of patient measurement, i.e. two weeks
  Comparison of the time to the first detection of atrial fibrillation or other arrhythmia when considering PPG-triggered ECG measurements or when considering the scheduled ECG measurements.
Evaluation of the accuracy of automatic ECG analysis algorithms when comparing with manual annotations by a cardiologist. | Duration of patient measurement, i.e. two weeks
  The automated assessment done for the 30-second ECG recordings is compared with the visual assessment to calculate the sensitivity and specificity for each rhythm category.

CONTACTS AND LOCATIONS:
Overall Officials: Vesa Virtanen, PhD (med), Principal Investigator — Heart Hospital of Tampere University Hospital
Locations (1):
- Tampere Heart Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No